CLINICAL TRIAL: NCT01861587
Title: Evaluation of the Effectiveness of tDCS in the Management of Perioperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: HR18682
Record Dates: First submitted 2012-04-26; First posted 2013-05-23 (Estimated); Results first posted 2018-07-10 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (2):
- Real tDCS:Active Comparator (Experimental): For Real tDCS, stimulation will be delivered in 20-minute-sessions using 2mA current. The anode will be placed over left BA9 or the motor cortex corresponding with the painful area (if applicable). The cathode will be placed over right BA43 (for GI pain) or right BA9 (located via the international 10-20 EEG system).
  Interventions: Device: tDCS
- Sham tDCS: Sham Comparator (Experimental): For sham tDCS, the device will be turned on for 30 seconds and then turned off for the duration of the 20-minute session.
  Interventions: Device: tDCS

INTERVENTIONS:
Device: tDCS — 20 minutes of either real or sham stimulation

SUMMARY:
The purpose of this study is to determine whether a new medical technology can help reduce post-operative pain. The new technology is called Transcranial Direct Current Stimulation.

DETAILED DESCRIPTION:
This study aims to evaluate the effectiveness of transcranial direct current stimulation (tDCS) in the management of postoperative pain. Specifically, this study will determine whether patients undergoing any type of inpatient surgical procedure that routinely requires at least a 1-day inpatient stay post-operatively will report less pain and use less opioid analgesics following a series of 20-minute sessions of tDCS (compared to sham tDCS) delivered up to twice per day post-operatively. In addition to comparing the effects of real tDCS to sham tDCS, the present study will evaluate the interaction of dose (number and frequency of tDCS sessions) and surgery type.

ELIGIBILITY:
Inclusion Criteria:

* 18 years-75 years of age
* surgery at Medical University of South Carolina
* at least 2 days of post-operative stay

Exclusion Criteria:

* history of seizures or epilepsy
* family history of seizures
* taking any medications shown to lower seizure threshold
* metal implants above the waist
* pregnant
* brain tumors or lesions
* pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Borckardt, Ph.D., Principal Investigator — Medical University of South Carolina
Locations (1):
- Brain Stimulation Laboratory, Institute of Psychiatry, Charleston, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator
Started | 14 | 13
Completed | 14 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator | Total
Number analyzed (Participants) | 14 | 13 | 27
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (2.1) | 59.4 (2.1) | 59.4 (2.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 8 | 17
  Male | 5 | 5 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 11 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 14 | 13 | 27

OUTCOME MEASURES:

1. Primary Outcome: Patient Controlled Analgesia (PCA) Hydromorphone Usage
Description: The PCA pump usage was downloaded from the PCA pump after discharge from the hospital.
Time Frame: Participants were followed for the duration of hospital stay, an average of 48 hours.
Measure: Mean (Standard Deviation); unit: milligrams of hydromorphone
Groups:
- Real tDCS:Active Comparator: tDCS: 20 minutes of stimulation at 2mA.
- Sham tDCS: Sham Comparator: For Sham tDCS, the stimulator was turned off automatically after 45 seconds.
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator
Number analyzed (Participants) | 14 | 13
milligrams of hydromorphone | 12.6 (9.9) | 16.5 (12.7)

2. Primary Outcome: Average Pain at Least
Description: To assess each participant's average pain at it's least in the past 24 hours, The Brief Pain Inventory (BPI)-short form will be administered. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their average pain at it's least in the past 24 hours using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: Baseline and Discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator
Number analyzed (Participants) | 14 | 13
units on a scale
  Baseline | 4.5 (2.5) | 3.5 (1.6)
  Discharge | 3.2 (2.2) | 3.5 (1.6)

3. Primary Outcome: Average Pain at Worst
Description: To assess each participant's average pain at it's worst in the past 24 hours at Baseline, The Brief Pain Inventory (BPI)-short form will be administered. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their average pain at it's worst in the past 24 hours using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: Baseline Only
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator
Number analyzed (Participants) | 14 | 13
units on a scale | 8.9 (1.2) | 8.0 (2.4)

4. Primary Outcome: Average Pain
Description: To assess each participant's pain on average in the past 24 hours at Baseline, The Brief Pain Inventory (BPI)-short form will be administered. The BPI rapidly assesses the severity of pain and its impact on functioning and has been widely used in both research and clinical settings. Participants rate their pain on average in the past 24 hours using a 0-10 numerical rating scale, where 0=no pain and 10=extreme pain.
Time Frame: Baseline Only
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Real tDCS: Real tDCS includes 20 minutes of stimulation at 2mA.
- Sham tDCS: For sham tDCS, the stimulator was turned off automatically after 45 seconds.
Arm/Group | Real tDCS | Sham tDCS
Number analyzed (Participants) | 14 | 13
units on a scale | 7.0 (1.5) | 6.3 (1.4)

ADVERSE EVENTS:
Time Frame: 2 Days
Arm/Group | Real tDCS:Active Comparator | Sham tDCS: Sham Comparator
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 0/14 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No